CLINICAL TRIAL: NCT04718610
Title: Effects of Vagus Nerve Osteopathic Stimulations on Heart Rate Variability of Cancer Patients
Brief Title: Heart Rate Variability, Vagus Nerve and Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Heart rate measurement error
Sponsor: Centre Hospitalier Henri Duffaut - Avignon (Other)
Collaborators: Institut de Formation en Ostéopathie du Grand Avignon (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSTEOCAN
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer; Colorectal Cancer; Multiple Myeloma; Non Hodgkin Lymphoma
Keywords: Cancer; Vagus nerve stimulation; Heart rate variability; Osteopathy
MeSH Terms: conditions — Lung Neoplasms; Colorectal Neoplasms; Multiple Myeloma; Lymphoma, Non-Hodgkin; Neoplasms

STUDY DESIGN:
Intervention Model Description: For each cancer type, 30 patients will be included. These patients will be randomized into two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients will receive only caner treatment. No osteopathic treatment.
  Interventions: Biological: CRP assessment; Behavioral: QLQ-C30 questionnaire
- Osteopathic intervention (Experimental): Patients will receive cancer treatment associated with osteopathic intervention
  Interventions: Other: Osteopathic intervention; Biological: CRP assessment; Behavioral: QLQ-C30 questionnaire

INTERVENTIONS:
Other: Osteopathic intervention — Nerve vagus stimulation
  Arms: Osteopathic intervention
Biological: CRP assessment — Blood CRP will be assessed during trial
Behavioral: QLQ-C30 questionnaire — Completion of QLQ-C30

SUMMARY:
In France, new cancer cases keep on increasing with around 150 000 deaths yearly. Cancer therapy research is constantly evolving. Indeed, several studies explore new treatments or their combination with conventional cancer treatments. But, at the same time, complementary and alternative medicines, as osteopathy, remain little explored upon their role in the combination with conventional therapy.

Several studies showed indirect interaction between vagus nerve and cancer. Firstly, vagus nerve regulates homeostasis and immunity by reducing systemic inflammation while maintaining local inflammation and antitumor effects. Secondly, vagus nerve stimulation increases Heart Rate Variability (HRV). Moreover, a higher HRV is associated with an improvement of vital prognosis in cancer patients. Vagus nerve could be stimulated by noninvasive osteopathic manipulations.

This prospective, monocentric and randomized study is a collaboration between the Centre Hospitalier d'Avignon and the Institut de Formation en Ostéopathie du Grand Avignon. It focuses on using noninvasive osteopathic mobilizations to stimulate vagus nerve. Indeed, this study aims to evaluate effects of vagus nerve osteopathic stimulations on HRV in patients with lung cancer, colorectal cancer, Non Hodgkin Lymphoma or Multiple Myeloma. More specifically, this study will tell us whether vagus nerve noninvasive osteopathic stimulations induce increase of HRV associated with a decrease of systemic inflammation and an improvement of patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient with lung cancer or colorectal cancer or Non Hodgkin Lymphoma or Multiple Myeloma (Stade I à IV)
* No previous treatment
* HRV < 70 ms
* No osteopathic contraindication

Exclusion Criteria:

* Vagotomy
* Heart arrhythmia
* Cancer recurrence
* Consumption of coffee or tabac within 2 hours prior osteopathic treatment
* Consumption of alcohol within 24 hours prior osteopathic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Change of Heart Rate Variability measured by SDNN (Standard Deviation of all NN intervals) from baseline to the end of osteopathic treatment | up to 84 days
  To assess the effect of vagus nerve osteopathic stimulations on Heart Rate Variability

SECONDARY OUTCOMES:
Serum concentration of C-Reactive Protein | up to 84 days
  To assess the effect of vagus nerve osteopathic stimulations on systemic inflammatory
Time to definitive improvement in global health status / QoL | up to 84 days
  To assess the effect of vagus nerve osteopathic stimulations on health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Borhane SLAMA, MD, Principal Investigator — Centre Hospitalier Henri Duffaut - Avignon
Locations (1):
- Centre Hospitalier Henri Duffaut, Avignon, France

IPD SHARING:
Plan to Share IPD: No